CLINICAL TRIAL: NCT04231773
Title: The Effect of Inhaled Nitric Oxide on Maximal Oxygen Consumption During Exercise in Hypoxia
Acronym: iNO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Pro00092939
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2022-07

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia | interventions — Nitric Oxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 12.1% Oxygen and Inhaled Nitric Oxide (Experimental): Moderate level of hypoxia (12.1% Oxygen) and Inhaled Nitric Oxide (40 ppm)
  Interventions: Drug: Nitric Oxide
- 12.1 % Oxygen Placebo (Placebo Comparator): Moderate level of hypoxia (12.1 % Oxygen) and Placebo (0 ppm Nitric Oxide)
  Interventions: Drug: Placebo
- 13.6 % Oxygen and Inhaled Nitric Oxide (Experimental): Severe level of hypoxia (13.6% Oxygen) and Inhaled Nitric Oxide (40 ppm)
  Interventions: Drug: Nitric Oxide
- 13.6 % Oxygen and Placebo (Placebo Comparator): Severe level of hypoxia (13.6% Oxygen) and Placebo (0 ppm Nitric Oxide)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nitric Oxide — 40 parts per million dosage
  Other Names: iNO
  Arms: 12.1% Oxygen and Inhaled Nitric Oxide; 13.6 % Oxygen and Inhaled Nitric Oxide
Drug: Placebo — Inhaled placebo. Device connected to same delivery system, but does not deliver nitric oxide.
  Other Names: Hypoxic Placebo
  Arms: 12.1 % Oxygen Placebo; 13.6 % Oxygen and Placebo

SUMMARY:
During exercise in conditions of low oxygen (termed hypoxia), such as mountaineering at high altitudes, the lung blood vessels constrict in an attempt to protect the body from the negative effects of hypoxia. It appears that this blood vessel constriction may limit the heart to pump blood during heavy exercise, leading to reductions in exercise performance. Inhaled nitric oxide is a drug that is known to relax the lung blood vessels. Inhaled nitric oxide has been used to relax lung blood vessels and improve exercise capacity in patients with chronic disease. It is unknown if similar improvements would be observed during exercise in healthy individuals when exposed to low levels of oxygen. The goal of this study is to determine if inhaled nitric oxide can relax the lung blood vessels and improve the heart's pumping ability during exercise in low oxygen conditions. Further, the investigators will determine if these improvements in lung blood vessel and heart function increase exercise performance. Participants will complete 6 sessions over a three week period where they will perform exercise challenges while breathing low levels of oxygen with and without inhaled nitric oxide. The low oxygen conditions will be comparable to being at an altitude of 14,000-17,000 feet. 17,000 feet would be equivalent to standing on the summit of King Peak in the Yukon (the 4th tallest mountain in Canada).

DETAILED DESCRIPTION:
Background

During exercise in hypoxic conditions, maximal exercise capacity, as determined by maximal oxygen uptake (V̇O2max), is reduced progressively as inspired oxygen tension falls. It is generally assumed that this reduction in V̇O2max results entirely from a reduction in arterial oxygen content. However, previous work in severe cases of hypoxia have demonstrated a larger than expected reduction in V̇O2max. Further, the hypoxia-induced impairment in V̇O2max could not be explained entirely by the reduced inspired O2 tension and suggest that other mechanisms contribute to the drop in V̇O2max. Previous research showed that impaired pulmonary gas-exchange and reduced peak cardiac output, in addition to the reduced arterial oxygen content, were key contributors to the impaired V̇O2max in severe hypoxia (10.5% inspired oxygen). The reason for the gas-exchange impairment and reduced cardiac output is currently unclear, however, it has been hypothesized that hypoxic pulmonary vasoconstriction (HPV) may increase pulmonary vascular resistance and pulmonary artery pressure during very heavy exercise. HPV-mediated increases in pulmonary vascular resistance would increase right heart work and potentially impair the pumping capacity of the heart, leading to a reduction in stroke volume and, ultimately, cardiac output. HPV has been detected, even in mild hypoxia (15-18% inspired oxygen), in healthy humans. Inhaled nitric oxide (iNO) is a selective pulmonary vasodilator and has been shown to reduce pulmonary vascular resistance during exercise in patients with pulmonary vascular dysfunction (i.e. chronic obstructive pulmonary disease). Further, iNO has been shown to release HPV in healthy individuals. If iNO can prevent HPV, this would mitigate the increase in pulmonary vascular resistance in moderate (~13.6% inspired oxygen) and more severe (~12.1% inspired oxygen) hypoxia and improve V̇O2max during hypoxic exercise. Therefore, we hypothesize that the iNO will improve V̇O2max during exercise in moderate and severe hypoxia, secondary to reduced pulmonary artery systolic pressure leading to increased stroke volume and peak cardiac output. Further, larger improvements in V̇O2max, with iNO, will be observed in severe hypoxia conditions, when compared to the iNO-mediated change in V̇O2max in moderate hypoxia. This would provide conclusive evidence that the pulmonary vasculature is a key contributor to reduced V̇O2max in both moderate and severe hypoxic conditions.

Trial Objectives

Purpose: To examine the effect of iNO on maximal oxygen consumption (V̇O2max) during exercise in hypoxia.

Hypothesis: Inhaled NO will improve V̇O2max during hypoxic exercise, secondary to increased stroke volume and peak cardiac output. A larger improvement in V̇O2max, with iNO, will be observed in more severe hypoxia conditions, when compared to the iNO-mediated change in V̇O2max in moderate hypoxia.

Study Design: Randomized double-blind cross-over design.

Study Protocol: Six sessions will be completed over a 3-week period in the following order: Day 1) Participant enrollment, medical history, standard pulmonary function (PFT) and cardiopulmonary exercise test (CPET) breathing normoxia (21% inspired oxygen). Days 2-5) Randomly-ordered experimental CPETs while either breathing A) moderate hypoxia (13.6% inspired oxygen), B) severe hypoxia (12.1% inspired oxygen), C) moderate hypoxia with 40 ppm iNO, and D) severe hypoxia with 40 ppm iNO. Day 6) Resting and exercise trials while breathing, normoxia, moderate and severe hypoxia, and moderate and severe hypoxia with iNO, with ultrasonography Doppler measurements to determine pulmonary arterial systolic pressure.

The hypoxia conditions will be comparable to being at an altitude of 14,000-17,000 feet. 17,000 feet would be equivalent to standing on the summit of King Peak in the Yukon (the 4th tallest mountain in Canada).

On Day 1, participants will complete the informed consent procedure, fill out a medical history questionnaire and be screened for exercise using a physical activity readiness questionnaire. They will undergo lung function and cardiopulmonary exercise testing on the same day. The participants will be spending approximately three hours in the laboratory on this testing day.

On days 2, 3, 4 & 5 the participants will breathe A) moderate hypoxia (13.6% inspired oxygen), B) severe hypoxia (12.1% inspired oxygen), C) moderate hypoxia with 40 ppm iNO, and D) severe hypoxia with 40 ppm iNO and have their blood flow/cardiac output and expired gas evaluated, and time to exhaustion determined in a standard cardiopulmonary exercise test. Prior to day two, the order of conditions will be block randomized to ensure both CPETs from one oxygen concentration (either 12.1 or 13.6 %) is completed before the second oxygen concentration condition is initiated.

On day 2, the participant will lie supine and be rested for 5 minutes. Their resting blood pressure will be determined using manual auscultation. Resting cardiac output will be evaluated using noninvasive impedance cardiography and oxygen saturation estimated with pulse oximetry. Ventilation will be measured from expired gas analysis. Following these measurements, the subject will begin to breathe one of the four experimental conditions (see above). Following a 5 minute wash-in period, ventilation, cardiac output and oxygen saturation recordings will be repeated. Participants will then perform a standard cardiopulmonary exercise test while continuing to breathe the normoxic air. The participants will be spending approximately three hours in the laboratory on this testing day.

Day 3, 4 & 5 will be identical to day 2 except, participants will breathe the other experimental conditions.

On Day 6 the subject will lie supine and be rested for 5 minutes to obtain supine baseline measurements. Following, participants will sit upright and baseline measurements will be recorded. Their resting systemic blood pressure will be determined using manual auscultation and pulmonary arterial systolic arterial pressure will be determine by cardiac ultrasound imaging. Resting cardiac output will be evaluated using noninvasive impedance cardiography. The resting measurements will be completed while breathing while breathing, normoxia, moderate and severe hypoxia, and moderate and severe hypoxia with iNO (order randomized). Participants will then completed short bouts of light exercise at a fixed intensity and all measurements will be repeated while breathing normoxia, moderate and severe hypoxia, and moderate and severe hypoxia with iNO (order randomized). The research participants will exercise at a light intensity for a total of ~25 minutes (5 minutes per conditions). For both the resting and exercise measurements, a 10-minute washout time will be given when switching between conditions.

Participant Duration: Each visit will take approximately 3 hours. The total time duration for each participant will be approximately 18 hours.

Intervention

Inhaled Nitric Oxide Intervention: Inhaled NO is a selective pulmonary vasodilator and has been shown to improve blood flow to well-ventilated lung areas (i.e. improve ventilation-perfusion matching) in conditions with elevated vascular tone. Inhaled NO has been previously shown to lower pulmonary artery pressure during exercise in lung disease patients, while not affecting systemic blood pressure. It is important to note that a selective pulmonary vasodilator will be used instead of an intravenously infused vasodilator (e.g. prostacyclin) to avoid systemic vasodilation, severe arterial hypotension and syncope 19-20. Consistent with previous work, a standard 40 ppm dose of inhaled NO will be administered using a non-rebreathing circuit.

Statistical analysis and Interpretation A 1-way repeated measures ANOVA will be used to evaluate the changes in V̇O2max with 1) moderate and severe hypoxia and, 2) moderate and severe hypoxia with iNO during exercise, when compared to placebo (normoxic condition). Should a main effect be found, a Tukey post-hoc t-test with be completed to locate the differences. Should iNO improve V̇O2max, then this would suggest that a hypoxic-mediated increase in pulmonary vascular resistance is a key contributor to impaired cardiac output during moderate and severe hypoxic exercise.

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers and less than 10 pack years smoking history
* Young healthy males and females with normal lung function and no known history of cardiopulmonary disease.

Exclusion Criteria:

* Individuals with significant cardiovascular, metabolic, neuromuscular or any other disease that could contribute to abnormal respiratory and cardiovascular responses to exercise will be excluded.
* Individuals with musculoskeletal injuries that prevent them from completing cycle ergometry exercise trials will be excluded.
* For safety reasons, pregnant females will be excluded.
* Participants currently on oral steroids (i.e. prednisone) or phosphodiesterase type 5 (PDE5) inhibitors will be excluded.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2021-12-04 (Actual); Study Completion 2021-12-04 (Actual)

PRIMARY OUTCOMES:
Exercise Capacity | Within 20-25 minutes post-dose
  Exercise capacity as determined by maximal oxygen consumption (V̇O2max)

SECONDARY OUTCOMES:
Cardiac Output | Within 20-25 minutes post-dose
  Cardiac output as determined by impedance cardiography.
Pulmonary artery pressure | Within 20-25 minutes post-dose
  Pulmonary artery systolic pressure at rest and during exercise determined by echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Micahel Stickland, PhD, Principal Investigator — University of Alberta
Locations (1):
- Clinical Physiology Laboratory, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No